CLINICAL TRIAL: NCT04667819
Title: Clinical Efficacy of Wireless Micropump in Dry Eye Patients
Brief Title: Wireless Micropump in Dry Eye Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Collaborators: Tianjin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202076
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Dry Eye
Keywords: micropump; dry eye; sodium hyaluronate
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sodium hyaluronate (Experimental): Sodium hyaluronate has become a novel and effective eye drop for the treatment of the dry eye. However, we design a special method of usage of sodium hyaluronate in dry eye patients.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Drug: Sodium Hyaluronate — We usage a special type of anterior eye drug delivery system to conduct the transmission of sodium hyaluronate in dry eye patients.

SUMMARY:
The purpose of this study is to carry out a trial to get more convincing and valuable results of the wireless micropump in dry eye patients and compare the outcomes before and after eye drops usage. The investigators hope to investigate the micropump comprehensively, including the comparison of tear film break-up time, corneal epithelium defect percentage, and tear film thickness. To meet the demands of a trial, all the examination equipment should be the same for each patient, and this will limit the variations within a study.

DETAILED DESCRIPTION:
The purpose of this study is to carry out a trial to get more convincing and valuable results of the wireless micropump in dry eye patients and compare the outcomes before and after eye drops usage. The investigators hope to investigate the micropump comprehensively, including the comparison of tear film break-up time, corneal epithelium defect percentage, and tear film thickness. To meet the demands of a trial, all the examination equipment and methods should be the same for each patient, and this will limit the variations within a study.

ELIGIBILITY:
Inclusion Criteria:

* elimination of serious mental and psychological diseases;
* be accompanied by a parent or guardian who is able to give informed consent as demonstrated by signing a record of informed consent;
* be willing to comply with the clinical trial visit schedule as directed by the investigator;
* at baseline, be within the age range of 18 to 80 years old inclusive;
* BCVA≥1.0 of both eyes for each patient;
* dry eye test is BUT<5s and or Schimer test<5mm/5min；
* without other ophthalmic diseases;

Exclusion Criteria:

* At the same time, patients with other eye diseases (such as glaucoma, corneal opacity, uveitis, etc.) were diagnosed;
* serious mental and psychological diseases;
* history of refractive surgery;
* nystagmus or failure to cooperate;
* history of intraocular surgery;
* patients with systemic diseases (such as diabetes, hypertension, heart disease, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
tear film break-up time | change from baseline with OCCULUS at 6 months
  change before and after sodium hyaluronate with OCCULUS
tear film thickness | change from baseline with OCCULUS at 6 months
  change before and after sodium hyaluronate with OCCULUS
corneal epithelium defect percentage | change from baseline with OCCULUS at 6 months
  change before and after sodium hyaluronate with OCCULUS

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Director — Tianjin Eye Hospital; Xuexin Duan, professor, Principal Investigator — Tianjin University
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Resto PJ, Berthier E, Beebe DJ, Williams JC. An inertia enhanced passive pumping mechanism for fluid flow in microfluidic devices. Lab Chip. 2012 Jun 21;12(12):2221-8. doi: 10.1039/c2lc20858j. Epub 2012 Mar 23. PMID 22441561
- [Result] Kamal T, Watkins R, Cen Z, Rubinstein J, Kong G, Lee WM. Design and fabrication of a passive droplet dispenser for portable high resolution imaging system. Sci Rep. 2017 Jan 27;7:41482. doi: 10.1038/srep41482. PMID 28128365
- [Result] Kwon JW, Kim JS, Choi SB, Lee JH, Wee WR. Experimental study of an automated system for the delivery of eyedrops using a microinfusion pump. Am J Ophthalmol. 2005 Mar;139(3):547-9. doi: 10.1016/j.ajo.2004.08.051. PMID 15767073
- [Result] Huang PH, Nama N, Mao Z, Li P, Rufo J, Chen Y, Xie Y, Wei CH, Wang L, Huang TJ. A reliable and programmable acoustofluidic pump powered by oscillating sharp-edge structures. Lab Chip. 2014 Nov 21;14(22):4319-23. doi: 10.1039/c4lc00806e. PMID 25188786
- [Result] Wu Z, Cai H, Ao Z, Nunez A, Liu H, Bondesson M, Guo S, Guo F. A Digital Acoustofluidic Pump Powered by Localized Fluid-Substrate Interactions. Anal Chem. 2019 Jun 4;91(11):7097-7103. doi: 10.1021/acs.analchem.9b00069. Epub 2019 May 14. PMID 31083981